CLINICAL TRIAL: NCT03852784
Title: Osteoarticular Infections With Pneumococcal
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, clinical reserach assistant, Hospices Civils de Lyon
Other Study IDs: 19-074
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Bone and Joint Infection
Keywords: Bone and Joint Infection; Streptococcus peumoniae

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bone and joint infection with Streptococcus peumoniae: Patients having had an osteoarticular infection with Streptococcus peumoniae
  Interventions: Other: Bone and joint infection with Streptococcus peumoniae

INTERVENTIONS:
Other: Bone and joint infection with Streptococcus peumoniae — description of the osteoarticular infection with Streptococcus peumoniae

SUMMARY:
Osteoarticular infections at pneumococcal are rare, potentially serious and remain under diagnosed. They represent 3 at 10% of the arthritis septic in the literature. 190 cases have been published of 1965 at 2003. They represent 0.3% at 0.6% of the bacteraemia at Streptococcus peumoniae.

ELIGIBILITY:
Inclusion Criteria:

* patients having had a bone and joint infection with S pneumoniae, with or without device.

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having had a bone and joint infection with S pneumoniae, with or without device managed at the Croix-Rousse hospital
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Description and rate of bone or joint infection with S. pneumoniae | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Description of the type of infection due to S. pneumoniae : patients and type of implant, profile of the bacterium associated in the infection, medical and chirurgical treatment

SECONDARY OUTCOMES:
Rate of Treatment Failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Md,PhD, Study Director — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr/